CLINICAL TRIAL: NCT03447834
Title: Selective Intracoronary Hypothermia in Patients With ST-elevation Myocardial Infarction to Reduce Infarct Size
Brief Title: EUROpean Intracoronary Cooling Evaluation in Patients With ST-elevation Myocardial Infarction.
Acronym: EURO-ICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Abbott (Industry); Golden Jubilee National Hospital (Other Government); Onze Lieve Vrouwziekenhuis Aalst (Other); Rigshospitalet, Denmark (Other); Örebro University, Sweden (Other); Skane University Hospital (Other); University of Belgrade (Other); Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nico Pijls, N.H.J Pijls, MD, PhD, Professor of Cardiology, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EURO-ICE
Record Dates: First submitted 2018-02-02; First posted 2018-02-27 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Acute Myocardial Infarction; Reperfusion Injury
Keywords: intracoronary cooling
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 fashion to either routine PPCI (control arm) or intracoronary hypothermia in addition to PPCI (hypothermia arm). For the patients randomized to intracoronary hypothermia will follow the steps below.
  For the routine PPCI a regular guidewire will be advanced across the occlusion followed by pre-dilatation and/or (direct) stenting according to the operator's preference.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective intracoronary hypothermia + PPCI (Experimental): Patients will be eligible for this study if they are admitted for acute anterior wall ST-elevation myocardial infarction with total ST-segment deviation of at least 5 mm. If the patient has TIMI grade flow 0 or 1, the experimental arm will be treated by selective intracoronary hypothermia just before and after reperfusion, in addition to routine PPCI.
  Interventions: Other: Selective intracoronary hypothermia + PPCI
- Standard PPCI (Other): The control group will receive routine PPCI.
  Interventions: Other: Standard PPCI

INTERVENTIONS:
Other: Selective intracoronary hypothermia + PPCI — Selective intracoronary hypothermia is a new technique, recently tested for safety and feasibility in the SINTAMI trial. The procedure starts by advancing a guidewire beyond the occlusion in the culprit artery, followed by an OTWB that is inflated at the location of the occlusion, at a low pressure (4 atm), to prevent reperfusion. After that, a pressure/temperature wire will be advanced along the inflated OTWB and is placed in the distal coronary artery. Then the guidewire is removed and the lumen is used for infusion of saline. During the 'occlusion phase', saline at room temperature is infused for 10 minutes with distal coronary temperature 6-8°C below body temperature. After that, the balloon of the OTWB is deflated. Simultaneously, infusion is started with saline of 4°C, the so called 'reperfusion phase'. This is continued for 10 more minutes. After that, the OTWB can be retracted and the procedure can continue not different from routine PPCI.
  Other Names: Selective intracoronary hypothermia
  Arms: Selective intracoronary hypothermia + PPCI
Other: Standard PPCI — PPCI per routine
  Arms: Standard PPCI

SUMMARY:
In acute myocardial infarction, early restoration of epicardial and myocardial blood flow is of paramount importance to limit infarction size and create optimum conditions for favourable long-term outcome. Currently, restoration of epicardial blood flow is preferably and effectively obtained by primary percutaneous coronary intervention (PPCI). After opening the occluded artery, however, the reperfusion process itself causes damage to the myocardium, the so called "reperfusion injury". The phenomenon of reperfusion injury is incompletely understood and currently there is no established therapy for preventing it. Contributory factors are intramyocardial edema with compression of the microvasculature, oxidative stress, calcium overload, mitochondrial transition pore opening, micro embolization, neutrophil plugging and hyper contracture. This results in myocardial stunning, reperfusion arrhythmias and ongoing myocardial necrosis. There is general agreement that a large part of the cell death caused by myocardial reperfusion injury occurs during the first few minutes of reperfusion, and that early treatment is required to prevent it.

Myocardial hypothermia may attenuate the pathological mechanisms mentioned above. However, limited data are available on the beneficial effects of hypothermia to protect the myocardium from reperfusion damage. In animals, several studies demonstrated a protective effect of hypothermia on the infarction area. This effect was only noted when hypothermia was established before reperfusion. Hypothermia is therefore thought to attenuate several damaging acute reperfusion processes such as oxidative stress, release of cytokines and development of interstitial or cellular edema. Furthermore, it has been shown that induced hypothermia resulted in increased ATP-preservation in the ischemic myocardium compared to normothermia. The intracoronary use of hypothermia by infused cold saline in pigs was demonstrated to be safe by Otake et al. In their study, saline of 4°C was used without complications (such as vasospasm, hemodynamic instability or bradycardia) and it even attenuated ventricular arrhythmia significantly.

Studies in humans, however, have not been able to confirm this effect, which is believed to be mainly due to the fact that the therapeutic temperature could not reached before reperfusion in the majority of patients or not achieved at all. Furthermore, in these studies it was intended to induce total body hypothermia, which in turn may lead to systemic reactions such as shivering and enhanced adrenergic state often requiring sedatives, which may necessitate artificial ventilation.

In fact, up to now any attempt to achieve therapeutic myocardial hypothermia in humans with myocardial infarction, is fundamentally limited because of four reasons:

1. Inability to cool the myocardium timely, i.e. before reperfusion
2. Inability to cool the diseased myocardium selectively
3. Inability to achieve an adequate decrease of temperature quick enough
4. Inability to achieve an adequate decrease of temperature large enough

Consequently, every attempt to achieve effective hypothermia in ST-segment myocardial infarction in humans has been severely hampered and was inadequate. In the last two years, the investigators have developed a methodology overcoming all of the limitations mentioned above. At first, the investigators have tested that methodology in isolated beating pig hearts with coronary artery occlusion and next, the investigators have tested the safety and feasibility of this methodology in humans.

Therefore, the time has come to perform a proof-of-principle study in humans, which is the subject of this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Acute anterior wall ST-elevation myocardial infarction
* Total ST-segment deviation of at least 5 mm
* Presenting within 6 hours after onset of complaints
* TIMI 0 or 1 flow in the LAD
* Hemodynamically stable and in an acceptable clinical condition
* Able to give informed consent

Exclusion Criteria:

* Age <18 year or >80 year
* Cardiogenic shock or hemodynamically unstable patients
* Patients with previous myocardial infarction in the culprit artery of with previous bypass surgery
* Very tortuous or calcified coronary arteries
* Complex or long-lasting primary PCI expected
* Severe concomitant disease or conditions with a life expectancy of less than one year
* Inability to understand and give informed consent
* Known contra-indication for MRI
* Pregnancy
* Severe conduction disturbances necessitating implantation of temporary pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint- Infarct size | From date of randomization until the date of the MRI made after 3 months
  The primary endpoint is the final infarct size (expressed in % of left ventricular mass) on MRI, made 3 months after the infarction revealed by late gadolinium enhancement.

SECONDARY OUTCOMES:
Secondary endpoint, composite of all-cause mortality and hospitalization for heart failure at 3 | From date of randomization until 3 months later
  Composite of all-cause mortality and hospitalization for heart failure at 3 months
Secondary endpoint, composite of all-cause mortality and hospitalization for heart failure at 1 year | From date of randomization until 1 year later
  Composite of all-cause mortality and hospitalization for heart failure at 1 year
Secondary endpoint, all-cause mortality at 3 months | From date of randomization until 3 months later
  All-cause mortality at 3 months
Secondary endpoint, all-cause mortality at 1 year | From date of randomization until 1 year later
  All-cause mortality at 1 year
Secondary endpoint, hospitalization for heart failure at 3 months | From date of randomization until 3 months later
  Hospitalization for heart failure at 3 months
Secondary endpoint, hospitalization for heart failure at 1 year | From date of randomization until 1 year later
  Hospitalization for heart failure at 1 year
Secondary endpoint, cardiac death at 3 months | From date of randomization until 3 months later
  Cardiac death at 3 months
Secondary endpoint, cardiac death at 1 year | From date of randomization until 1 year later
  Cardiac death at 1 year
Secondary endpoint, peak value of high-sensitivity troponin T (hs-TnT) | From date of randomization until 1 week later
  Peak value of high-sensitivity troponin T (hs-TnT)
Secondary endpoint, peak value of creatine kinase (CK) | From date of randomization until 1 week later
  Peak value of creatine kinase (CK)
Secondary endpoint, peak value of creatine kinase-MB mass (CK-MB) | From date of randomization until 1 week later
  Peak value of creatine kinase-MB mass (CK-MB)
Secondary endpoint, echocardiography outcome | From date of randomization until 3 months later
  Left ventricular ejection fraction measured by echocardiography (biplane Simpson's method) at 3 months
Secondary endpoint, echocardiography outcome | From date of randomization until 1 year later
  Left ventricular ejection fraction measured by echocardiography (biplane Simpson's method) at 1 year
Secondary endpoint, echocardiography outcome | From date of randomization until 3 months later
  Wall motion score index (WMSI) by echocardiography at 3 months
Secondary endpoint, echocardiography outcome | From date of randomization until 1 year later
  Wall motion score index (WMSI) by echocardiography at 1 year
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  First pass microvascular obstruction extent (FP MVO); NB first pass will be acquired in 3 SAX levels to provide an index of %LV FP MVO
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Early MVO extent (% of LV) on 1 min post-gadolinium contrast enhanced MRI, adjusted for area at-risk
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Late MVO (presence / absence) on LGE
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Initial infarct size (LGE)
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Initial MSI (area-at-risk minus initial infarct size/area-at-risk)
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Left ventricular end-diastolic volume index (LVEDVI)
Secondary endpoint, MRI efficacy at baseline | From date of randomization until 5-7 days later; baseline MRI
  Left ventricular end-systolic volume index (LVESVI)
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Left ventricular global longitudinal strain
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Left ventricular circumferential strain (mid-LV)
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Left ventricular ejection fraction (LVEF)
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Systolic wall thickening in the culprit artery territory
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Wall motion score index (WMSI)
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Myocardial haemorrhage (presence/absence)
Secondary endpoint, MRI outcome at baseline | From date of randomization until 5-7 days later; baseline MRI
  Myocardial haemorrhage extent (% of LV)
Secondary endpoint, MRI outcome at follow-up | From date of randomization until 3 months later; follow-up MRI
  Final myocardial salvage index (area-at-risk minus final infarct size/area-at-risk)
Secondary endpoint, MRI outcome at follow-up | From date of randomization until 3 months later; follow-up MRI
  Change in infarct size 3 months after procedure (LGE at baseline minus LGE at 3 months)
Secondary endpoint, MRI outcome at follow-up | From date of randomization until 3 months later; follow-up MRI
  Final left ventricular end-diastolic volume index (LVEDVI)
Secondary endpoint, MRI outcome at follow-up | From date of randomization until 3 months later; follow-up MRI
  Final left ventricular end-systolic volume index (LVESVI)
Secondary endpoint, MRI outcome at follow-up | From date of randomization until 3 months later; follow-up MRI
  Final left ventricular ejection fraction (LVEF)
Secondary endpoint, MRI outcome at follow-up | From date of randomization until 3 months later; follow-up MRI
  Final left ventricular global longitudinal strain
Secondary endpoint, MRI outcome at follow-up | From date of randomization until 3 months later; follow-up MRI
  Final left ventricular circumferential strain (mid-LV)
Secondary endpoint, MRI outcome, difference between baseline and follow-up | From date of randomization until 3 months later; follow-up MRI
  Change from baseline left ventricular end-diastolic volume index (LVEDVI)
Secondary endpoint, MRI outcome, difference between baseline and follow-up | From date of randomization until 3 months later; follow-up MRI
  Change from baseline left ventricular end-systolic volume index (LVESVI)
Secondary endpoint, MRI outcome, difference between baseline and follow-up | From date of randomization until 3 months later; follow-up MRI
  Change from baseline left ventricular ejection fraction (LVEF)
Secondary endpoint, MRI outcome, difference between baseline and follow-up | From date of randomization until 3 months later; follow-up MRI
  Change in left ventricular global longitudinal strain
Secondary endpoint, MRI outcome, difference between baseline and follow-up | From date of randomization until 3 months later; follow-up MRI
  Change in left ventricular circumferential strain (mid-LV)

OTHER OUTCOMES:
Pre-specified subgroup analyses, between the hypothermia and control arm, as well as within each arm, as appropriate. | From date of randomization of last patient until 1 year later
  Comparison of outcomes by baseline features including diabetes status, sex, age and geographic location.
Pre-specified subgroup analyses, between the hypothermia and control arm, as well as within each arm, as appropriate. | From date of randomization of last patient until 1 year later
  Comparison of outcomes by lesion location (proximal versus mid LAD)
Pre-specified subgroup analyses, between the hypothermia and control arm, as well as within each arm, as appropriate. | From date of randomization of last patient until 1 year later
  Comparison of outcomes by TIMI grade flow (0 versus 1)
Pre-specified subgroup analyses, between the hypothermia and control arm, as well as within each arm, as appropriate. | From date of randomization of last patient until 1 year later
  Comparison of outcomes by achieved decrease in distal temperature (using median of cohort for threshold)

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El Farissi M, Pijls NHJ, Good R, Engstrom T, Keeble TR, Beleslin B, De Bruyne B, Frobert O, Erlinge D, Teeuwen K, Eerdekens R, Demandt JPA, Mangion K, Lonborg J, Setz-Pels W, Karamasis G, Wijnbergen I, Vlaar PJ, de Vos A, Brueren GR, Oldroyd K, Berry C, Tonino PAL, Van't Veer M, Otterspoor LC. A randomised trial of selective intracoronary hypothermia during primary PCI. EuroIntervention. 2024 Jun 17;20(12):e740-e749. doi: 10.4244/EIJ-D-23-01042. PMID 38887884
- [Derived] El Farissi M, Good R, Engstrom T, Oldroyd KG, Karamasis GV, Vlaar PJ, Lonborg JT, Teeuwen K, Keeble TR, Mangion K, De Bruyne B, Frobert O, De Vos A, Zwart B, Snijder RJR, Brueren GRG, Palmers PJ, Wijnbergen IF, Berry C, Tonino PAL, Otterspoor LC, Pijls NHJ. Safety of Selective Intracoronary Hypothermia During Primary Percutaneous Coronary Intervention in Patients With Anterior STEMI. JACC Cardiovasc Interv. 2021 Sep 27;14(18):2047-2055. doi: 10.1016/j.jcin.2021.06.009. Epub 2021 Aug 25. PMID 34454860